CLINICAL TRIAL: NCT03001635
Title: The Impact of Oxytocin Administration on Short and Long Term Prognosis in Patients Undergoing ST Elevation Myocardial Infarction
Brief Title: Role of Oxytocin in Myocardial Infarction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2629-15-SMC
Record Dates: First submitted 2016-12-14; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional treatment and oxytocin (Experimental): 26 patients admitted to the ICCU under a diagnosis of STEMI will receive treatment with oxytocin as an add on to the conventional treatment (e.g. primary PCI, aspirin, ADP receptor inhibitors, high dose statin, beta blockers & ACE inhibitors). At admission, a continuance infusion with oxytocin will be initiated for a time period of 6 hours. 10 units of oxytocin will be diluted in 1 liter of 0.9% normal saline. the infusion will start at a rate of 2.5 milliunits/min. dosage will be increased at a rate of 5 milliuinits/min every 30 min if there are no side effect, up to a maximum dosage of 30 milliunits/min.
  Interventions: Drug: Oxytocin
- conventional treatment only (Placebo Comparator): 26 patients admitted to the ICCU under a diagnosis of STEMI will receive the conventional treatment (e.g. primary PCI, aspirin, ADP receptor inhibitors, high dose statin, beta blockers & ACE inhibitors). On admission, an infusion of 0.9 normal saline will be stared as placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin — 26 patients will receive Oxytocin infusion for 6h while 26 will receive placebo. all other treatments will be the same and up to date with the current guidelines.
  Other Names: Pitocin
  Arms: conventional treatment and oxytocin
Drug: Placebos — 26 patients will receive 0.9% normal saline infusion for 6h as placebo
  Arms: conventional treatment only

SUMMARY:
60 patients admitted to this ICCU at the Sheba medical Center will be randomly divided in to 2 groups. one group will receive the conventional treatment while the second group will receive the conventional treatment plus oxytocin infusion for 48 hours. all participants will undergo echo and cMRI during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* current diagnosis of ST elevation myocardial infarction
* no previous episodes of acute coronary syndrome
* agreed to enter research

Exclusion Criteria:

* age < 18 years
* congestive heart failure (acute or chronic)
* cardiomyopathy
* life threatening arrhythmia at presentation
* previous LV dysfunction
* hypotension (systolic < 100mmHg, diastolic<50mmHg, 15% less than patients normal values)
* tachycardia - pulse > 100bpm
* bradycardia - pulse < 55 ppm
* killip 3 or 4 at presentation
* current use of nitrates
* pregnancy
* females - history of pathological GU bleeding
* inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
final infarction size | 1 week
  all patients will undergo an cMRI after 7 days

SECONDARY OUTCOMES:
Ejection fraction | 48 hours
  all patients will undergo echocardiography exam during the first 48 hours

OTHER OUTCOMES:
number on events with ventricular arrythmia | 48 hours
  all patients will be continually monitored for ventricular arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Anat Berkovitch, resident, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robinson KJ, Hazon N, Lonergan M, Pomeroy PP. Validation of an enzyme-linked immunoassay (ELISA) for plasma oxytocin in a novel mammal species reveals potential errors induced by sampling procedure. J Neurosci Methods. 2014 Apr 15;226:73-79. doi: 10.1016/j.jneumeth.2014.01.019. Epub 2014 Jan 28. PMID 24485867
- [Result] Danalache BA, Paquin J, Donghao W, Grygorczyk R, Moore JC, Mummery CL, Gutkowska J, Jankowski M. Nitric oxide signaling in oxytocin-mediated cardiomyogenesis. Stem Cells. 2007 Mar;25(3):679-88. doi: 10.1634/stemcells.2005-0610. Epub 2006 Nov 30. PMID 17138963
- [Result] Gutkowska J, Jankowski M. Oxytocin revisited: its role in cardiovascular regulation. J Neuroendocrinol. 2012 Apr;24(4):599-608. doi: 10.1111/j.1365-2826.2011.02235.x. PMID 21981277
- [Result] Jankowski M, Wang D, Hajjar F, Mukaddam-Daher S, McCann SM, Gutkowska J. Oxytocin and its receptors are synthesized in the rat vasculature. Proc Natl Acad Sci U S A. 2000 May 23;97(11):6207-11. doi: 10.1073/pnas.110137497. PMID 10811917
- [Result] Alizadeh AM, Faghihi M, Sadeghipour HR, Mohammadghasemi F, Imani A, Houshmand F, Khori V. Oxytocin protects rat heart against ischemia-reperfusion injury via pathway involving mitochondrial ATP-dependent potassium channel. Peptides. 2010 Jul;31(7):1341-5. doi: 10.1016/j.peptides.2010.04.012. Epub 2010 Apr 22. PMID 20417240
- [Result] Jankowski M, Hajjar F, Kawas SA, Mukaddam-Daher S, Hoffman G, McCann SM, Gutkowska J. Rat heart: a site of oxytocin production and action. Proc Natl Acad Sci U S A. 1998 Nov 24;95(24):14558-63. doi: 10.1073/pnas.95.24.14558. PMID 9826739
- [Result] Ondrejcakova M, Barancik M, Bartekova M, Ravingerova T, Jezova D. Prolonged oxytocin treatment in rats affects intracellular signaling and induces myocardial protection against infarction. Gen Physiol Biophys. 2012 Sep;31(3):261-70. doi: 10.4149/gpb_2012_030. PMID 23047939
- [Result] Jankowski M, Bissonauth V, Gao L, Gangal M, Wang D, Danalache B, Wang Y, Stoyanova E, Cloutier G, Blaise G, Gutkowska J. Anti-inflammatory effect of oxytocin in rat myocardial infarction. Basic Res Cardiol. 2010 Mar;105(2):205-18. doi: 10.1007/s00395-009-0076-5. Epub 2009 Dec 12. PMID 20012748
- [Result] Anvari MA, Imani A, Faghihi M, Karimian SM, Moghimian M, Khansari M. The administration of oxytocin during early reperfusion, dose-dependently protects the isolated male rat heart against ischemia/reperfusion injury. Eur J Pharmacol. 2012 May 5;682(1-3):137-41. doi: 10.1016/j.ejphar.2012.02.029. Epub 2012 Mar 3. PMID 22406244
- [Result] Authier S, Tanguay JF, Geoffroy P, Gauvin D, Bichot S, Ybarra N, Otis C, Troncy E. Cardiovascular effects of oxytocin infusion in a porcine model of myocardial infarct. J Cardiovasc Pharmacol. 2010 Jan;55(1):74-82. doi: 10.1097/FJC.0b013e3181c5e7d4. PMID 19858734